CLINICAL TRIAL: NCT04788901
Title: The Validity of In-game Performance Measurements or Scores as Indicators of Children's Emotional Regulation Abilities
Brief Title: Assessment of Emotion-regulation Skills in Game-based Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Associate Professor, Babes-Bolyai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1693/22.02.2021
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Emotional Problem
Keywords: emotional regulation; online therapeutic game; emotional regulation assessment
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online therapeutic game (Experimental): Participants in this group will have access to the evaluation module of the REThink game.
  Interventions: Other: REThink therapeutic game

INTERVENTIONS:
Other: REThink therapeutic game — REThink is a online therapeutic game developed by David and collaborators (2018), proved to be an efficient intervention to reduce emotional symptoms of children and adolescents.

SUMMARY:
The aim of the study is to investigate the validity of in-game scores as indicators for emotional regulation abilities in children and adolescence.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents between 10 and 14 years
* provided written parental consent

Exclusion Criteria:

* Intellectual disability or physical limitations precluded the use of the computer program
* Had a major mental health disorder

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Emotion-regulation | Pre-intervention (one day before the intervention)
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001). It is a 13-item on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities,
Strengths and difficulties | Pre-intervention (one day before the intervention)
  Strengths and Difficulties Questionnaire - child version (SDQ; Goodman, 1997). It is a 25-item on a three-point Liker scale, from 0 "not true" to 2 "certainly true" where lower scores represent an improvement or lack of problems.
Emotional symptoms | Pre-intervention (one day before the intervention)
  The Child Behavior Checklist for ages 6-18 (CBCL; Achenbach & Rescorla, 2001) is a parent-report of child emotional and behavioral problems. Each item is rated on a 3-point Likert-style scale ranging from 0 (not true) to 2 (very true or often true). The DSM-derived affective and anxiety scales and the anxious/depressed and withdrawn/depressed syndrome scales, respectively, will be used to assess emotional symptoms.
Emotion recognition | Pre-intervention (one day before the intervention)
  The Emotion Awareness Questionnaire (EAQ, Rieffe et al., 2008) is a 32-item questionnaire on a three-point Liker scale, from 0 "not true" to 2 "certainly true".
Compassion | Pre-intervention (one day before the intervention)
  Compassion Scale for Children (CSC, Nas & Sak, 2020) is a 20-items scale rated on a five points Likert scale from "Never" to "Always" where higher scores means higher levels of compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Derived] David OA, Tomoiaga C, Fodor LA. Gamified Assessment of the Emotion Regulation Abilities in Youth: Validation of the REThink Online System. Games Health J. 2024 Jun;13(3):184-191. doi: 10.1089/g4h.2023.0011. Epub 2024 Jan 24. PMID 38265781